CLINICAL TRIAL: NCT04091503
Title: Pilot Study to Evaluate the Safety, Tolerability and Effectiveness of Intranasal Administration of Temozolomide in Patients With Glioblastoma (Phase I)
Brief Title: Evaluate the Safety and Effectiveness of Intranasal Administration of Temozolomide in Patients With Glioblastoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Center Trials & Treatment Europe (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 7SQZ309D4W
Record Dates: First submitted 2019-09-08; First posted 2019-09-16 (Actual); Last update posted 2023-04-25 (Actual); Status verified 2023-04

CONDITIONS: Glioma, Malignant; Gliosarcoma; Astrocytoma of Brain
Keywords: TMZ; Temozolomide; Intranasal Administration; Nasal Spray; Intranasal Modified Temozolomide
MeSH Terms: conditions — Glioma; Gliosarcoma | interventions — Temozolomide

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Intranasal Modified Temozolomide 75 mg/M2 per day (Active Comparator): 75 mg/M2 per day Intranasal Modified Temozolomide administration of within 5 days per week (max: 30 days)
  Interventions: Drug: Intranasal Modified Temozolomide
- Intranasal Modified Temozolomide 150 mg/M2 per day (Active Comparator): 150 mg/M2 per day Intranasal Modified Temozolomide administration of within 5 days per week (max: 30 days)
  Interventions: Drug: Intranasal Modified Temozolomide
- Intranasal Modified Temozolomide 200 mg/M2 per day (Active Comparator): 200 mg/M2 per day Intranasal Modified Temozolomide administration of within 5 days per week (max: 30 days)
  Interventions: Drug: Intranasal Modified Temozolomide

INTERVENTIONS:
Drug: Intranasal Modified Temozolomide — Intranasally Modified Temozolomide is administered to patients at a dose of 75/150/200 mg / M2 for five days continuously. After the 5-day course, patients do not take treatment for two days, and they will be examined on an outpatient basis (blood tests, kidney and liver tests, visually mucous membranes of the mouth, nasal cavity, olfactory rapid tests, including the University of Pennsylvania test, etc.).
  After 30 days after the first intranasal administration of Modified Temozolomide (IM-TMZ), all patients undergo an MRI of the brain with perfusion and ultrasound of the abdominal cavity as an outpatient, after which the results are evaluated
  Other Names: Temozolomide; TMZ; IM-TMZ

SUMMARY:
The purpose of this pilot study is to determine the safety, tolerability, and the maximum tolerated dose intranasal administration of temozolomide (TMZ) as a single agent in Treatment on the patients with GBM.

Intranasal administration is a new method of treating brain tumours for the direct administration of drugs, inhibitors or viruses, with minimal involvement of the BBB. The investigators know the orally prescribed standard chemotherapy temozolomide (TMZ) is widely used to treat glioma tumours.

Received evidence of safety and efficacy in a full cycle of preclinical trials (on GLP Standart) and tests of calculated doses of intranasal administration of TMZ in healthy volunteers.

Intranasal administration of temozolomide is considered as GBM therapy, which provides direct access to a therapeutic dose of the drug into the brain (to the neoplastic process) with low toxicity

DETAILED DESCRIPTION:
The investigators are trying to evaluate a clinically potentially effective intranasal way of delivering TMZ to the brain, taking into account the anatomical structure of os ethmoidal.

The most important factor in the effectiveness of the drug is the achievement of an adequate amount of the active agent in its unbound state with albumin on the blood of a patient and the exposure time to the tumour process. Failure to comply with this requirement (difficulties in overcoming the BBB) was identified as the main obstacle to the successful treatment of all types of brain tumours. Translation to improved clinical outcomes in a patient with GBM has not yet been realized. The investigators will use modified temozolomide (without changing the chemical formula) to exclude as much as possible Anosmia, Hyposmia and other violation of the identification of odours with participants.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent signed
* 21 years or older
* Histologically confirmed the diagnosis of Grade 4 astrocytic tumour, which includes glioblastoma, giant cell glioblastoma, gliosarcoma, and glioblastoma with oligodendroglial components
* The availability of histological material for the possibility of revising histological verification
* IDH 1 Mutation and IDH2 Mutation are not taken into account when enrolling in that study
* MGMT promoter methylation MUST BE CONFIRMED
* Must have a Karnofsky performance status of ≥ 70% and the ability to use intranasal administration
* Sexually active fertile subjects (male and female) must agree to use accepted methods of contraception during the course of the study and for 3 months after the last intranasal administration of Temozolomide
* Female subjects of childbearing potential must have a negative pregnancy test at screening.
* Must be capable of understanding and complying with the protocol requirements

Exclusion Criteria:

* History of hypersensitivity to TMZ or any of its excipients
* The subject has had major surgery within 28 days prior to starting study treatment, or had non-water-tight dural closure during previous surgery, or has unhealed wounds from previous surgery
* The subject has inherited bleeding diathesis or coagulopathy with the risk of bleeding.
* The subject is pregnant or breastfeeding
* The subject suffered a stroke according to the results of the first MRI upon admission
* Anti-cancer Agents: Subjects who are currently receiving other anticancer agents are not eligible. Subjects must have fully recovered from the effects of prior chemotherapy (haematological and bone marrow suppression effects), generally at least 3 weeks from the most recent administration (6 weeks for nitrosoureas). Subjects may not have received more than 1 cycle of Irinotecan and Temozolomide as previous relapse therapy
* Subject is unable or unwilling to abide by the study protocol or cooperate fully with the investigator or designee

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2019-12-20 (Actual); Primary Completion 2022-09-21 (Actual); Study Completion 2022-10-28 (Actual)

PRIMARY OUTCOMES:
The randomized study to determine the safety of Intranasal Administration of modified Temozolomide. | up to 60 days (or withdrawal of consent or another discontinuation criterion) from date of randomization
  Incidence of Treatment-Emergent Adverse Events will be estimated by the number of participants with Glioblastoma or Gliosarcoma according to the NCI CTC (5.0) with adverse events (AE) in all cohorts.

SECONDARY OUTCOMES:
The maximum tolerated therapeutic dose (MTD) of modified Temozolomide for intranasal administration | up to 90 days (or withdrawal of consent or another discontinuation criterion) from date of randomization
  In the present study, the maximum dose of modified Temozolomide for intranasal administration is 200 mg / M2 a single daily intranasal administration in a course of 5 days. The frequency of adverse events, unacceptable toxicity, or haematological reactions is estimated on a scale the NCI CTCAE (v. 5.0)

OTHER OUTCOMES:
Percentage of Participants Alive 6 Months After Start of Treatment of Temozolomide for intranasal administration | 180 days
  Overall survival (OS) will be determined as the time in days from the start of treatment ( randomizations day ) to death due to any cause was estimated by the Kaplan-Meier method.
  If it was not known for certain that the participant to die, time will be censored at the last date the participant with GBM or Gliosarcomawas known to be alive, date of magnetic resonance imaging (MRI), etc, - assessment, which will be defined as the latest among the date of the last visit.
The effectiveness of intranasal administration of modified Temozolomide | up to 90 days (or withdrawal of consent or another discontinuation criterion) from date of randomization
  The effectiveness of the intranasal administration of modified Temozolomide will be evaluated by four MRIs with perfusion (first MRI performed one day before randomization day). The results of all MRI in dynamics will be appreciated by a consultation of radiologists.

CONTACTS AND LOCATIONS:
Locations (3):
- Central Contact, Banja Luka, Bosnia and Herzegovina
- Central Contact, Plovdiv, Bulgaria
- Central Contact, Tbilisi, Georgia

IPD SHARING:
Plan to Share IPD: No